CLINICAL TRIAL: NCT00171860
Title: A Study to Determine the Safety and Efficacy of Imatinib Mesylate in Patients With Idiopathic Hypereosinophilic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571ABE01
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Hypereosinophilic Syndrome
Keywords: Hypereosinophilic syndrome; Imatinib
MeSH Terms: conditions — Hypereosinophilic Syndrome | interventions — Imatinib Mesylate

ARMS (1):
- STI571 (Experimental)
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate
  Other Names: Gleevec/Glivec

SUMMARY:
The objectives of the study are:

1. Evaluation of the safety profile of imatinib mesylate in patients with idiopathic hypereosinophilic syndrome resistant or refractory to, or intolerant of, prednisone, hydroxyurea or interferon-alpha, or untreated patients carrying the Fip1L1-PDGFRA fusion protein.
2. Evaluation of the efficacy of imatinib mesylate in patients with idiopathic hypereosinophilic syndrome
3. Analysis of patient's blood samples for the detection of activated kinases.

ELIGIBILITY:
Inclusion Criteria:

Idiopathic hypereosinophilic syndromes are included provided they belong to one of the following categories:

1. previously treated and showing documented resistance or refractoriness to, or intolerance of, prednisone, hydroxyurea or interferon-alpha.
2. not previously treated but with documented Fip1L1-PDGFRA fusion protein

Exclusion Criteria:

* Other diseases associated with hypereosinophilia
* Serum creatinine, serum bilirubin, AST, ALT more than twice the upper normal limit.
* ECOG performance status >3

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-09; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Rate of complete and partial response and relapse

SECONDARY OUTCOMES:
Bone Marrow Analysis
Peripheral blood detection of Fip1L1-PDGFRA tyrosine kinase
Disease-Related Symptoms and Signs
Organ Involvement

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Leuven, Belgium